CLINICAL TRIAL: NCT02362711
Title: Phase3, Placebo Controlled, Randomized, Double-blinded, Long-Term, NSAID-Add-on, Clinical Trial of NPC-16 for Treatment of Dysmenorrhea
Brief Title: Efficacy and Safety, Long-Term Study of NPC-16 to Treat Dysmenorrhea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nobelpharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NPC-16-2
Record Dates: First submitted 2015-02-09; First posted 2015-02-13 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2015-02

CONDITIONS: Dysmenorrhea
MeSH Terms: conditions — Dysmenorrhea | interventions — Levonorgestrel; Ethinyl Estradiol; NPC 16

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- NPC-16 Standard Dosing Regimen Group (Experimental): Levonorgestrel 0.09mg, Ethinylestradiol 0.02mg
  Interventions: Drug: NPC-16 Standard Dosing Regimen Group
- NPC-16 Continuous Dosing Regimen Group (Experimental): Levonorgestrel 0.09mg, Ethinylestradiol 0.02mg
  Interventions: Drug: NPC-16 Continuous Dosing Regimen Group
- Placebo Group (Placebo Comparator): Placebo for NPC-16
  Interventions: Drug: Placebo Group

INTERVENTIONS:
Drug: NPC-16 Standard Dosing Regimen Group
  Other Names: Levonorgestrel 0.09mg, Ethinylestradiol 0.02mg
  Arms: NPC-16 Standard Dosing Regimen Group
Drug: NPC-16 Continuous Dosing Regimen Group
  Other Names: Levonorgestrel 0.09mg, Ethinylestradiol 0.02mg
  Arms: NPC-16 Continuous Dosing Regimen Group
Drug: Placebo Group
  Other Names: Placebo for NPC-16
  Arms: Placebo Group

SUMMARY:
The purpose of this long-term study is to determine whether NPC-16 is effective in the treatment of dysmenorrhea.

ELIGIBILITY:
Inclusion Criteria:

* dysmenorrhea

Exclusion Criteria:

* severe hepatopathy
* pregnant woman

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01-28 (Actual)

PRIMARY OUTCOMES:
Patient Response to Treatment for Dysmenorrhea, as Evaluated by Total Dysmenorrhea Score | 52 weeks

SECONDARY OUTCOMES:
Patient Response to Treatment for Dysmenorrhea, as Evaluated by Visual Analogue Scale (VAS) of Dysmenorrhea | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tasuku Harada, MD, PhD, Study Chair — Tottori University; Mikio Momoeda, MD, PhD, Study Chair — St. Luke's International Hospital